CLINICAL TRIAL: NCT01034241
Title: Effect of Different Protein Diets on Glucose and Insulin Metabolism and Substrate Partitioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nederlandse Zuivel Organisatie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MEC 08-3-072
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Insulin; Glucose Metabolism
Keywords: milk protein; overweight; insulin metabolism; substrate partitioning
MeSH Terms: conditions — Insulin Resistance; Overweight | interventions — Plant Proteins, Dietary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Experimental): Diet consists of 15% dairy protein and low Glycemic Index (GI < 40), 55 En% carbohydrates and 30 En% fat
  Interventions: Dietary Supplement: Control
- High dairy protein (Experimental): Diet consists of 25% dairy protein and low GI (GI < 40), 45 En% carbohydrates and 30 En% fat
  Interventions: Dietary Supplement: High dairy protein
- vegetable protein (Experimental): Diet consists of 15 En% vegetable protein and low GI (GI < 40), 55 En% carbohydrates and 30 En% fat
  Interventions: Dietary Supplement: vegetable protein
- High GI (Experimental): Diet consists of 15 En% dairy protein and high GI(GI > 60, 55 En% carbohydrates and 30 En% fat
  Interventions: Dietary Supplement: High GI

INTERVENTIONS:
Dietary Supplement: Control — Diet consists of 15 En% dairy protein and low GI, 55 En% carbohydrates and 30 En% fat
  Arms: Control
Dietary Supplement: High dairy protein — Diet consists of 25 En% dairy protein and low GI, 55 En% carbohydrates and 30 En% fat
  Arms: High dairy protein
Dietary Supplement: vegetable protein — Diet consists of 15 En% vegetable protein and low GI, 55 En% carbohydrates and 30 En% fat
  Arms: vegetable protein
Dietary Supplement: High GI — Diet consists of 15 En% dairy protein and high GI, 55 En% carbohydrates and 30 En% fat
  Arms: High GI

SUMMARY:
The purpose of this study is to determine whether different protein diets affects glucose and insulin metabolism and substrate partitioning.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-25 kg/m2 (lean)
* Gender: Male
* Age: <35 years
* Caucasian

Exclusion Criteria:

* Elevated fasting blood glucose level
* Lactose intolerant
* Diabetes Mellitus
* Hypertension (systolic/diastolic blood pressure)
* Hypotension (systolic/diastolic blood pressure)
* Cardiovascular diseases
* Asthma and other obstructive pulmonary diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Glucose and insulin metabolism (24 h) | 24 h

SECONDARY OUTCOMES:
Substrate partitioning and metabolic markers | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Wim Saris, Prof. Dr., Principal Investigator — Maastricht University

REFERENCES:
- [Derived] Munsters MJ, Geraedts MC, Saris WH. Effects of different protein and glycemic index diets on metabolic profiles and substrate partitioning in lean healthy males. Appl Physiol Nutr Metab. 2013 Nov;38(11):1107-14. doi: 10.1139/apnm-2012-0409. Epub 2013 Apr 25. PMID 24053517